CLINICAL TRIAL: NCT05144477
Title: Family-Authored ICU Diaries to Reduce Fear in Patients Experiencing a Cardiac Arrest (FAID Fear): A Pilot Intervention Study
Brief Title: Family-Authored ICU Diaries to Reduce Fear in Patients Experiencing a Cardiac Arrest (FAID Fear)
Acronym: FAID Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Talea M. Cornelius, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAT7681; P30AG064198 (NIH)
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Results first posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Cardiac Arrest; Post Traumatic Stress Syndrome
Keywords: Family Members; Couples; Partners; Fear; Fear of Exercise; Physical Activity
MeSH Terms: conditions — Heart Arrest; Combat Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAID Fear Intervention (Experimental): Family members of CA patients assigned to intervention will receive the ICU diary.
  Interventions: Behavioral: FAID Fear Intervention
- Control condition - Usual Care (No Intervention): Family members of CA patients assigned to usual care will not receive the ICU diary.

INTERVENTIONS:
Behavioral: FAID Fear Intervention — Participants will receive a hard-cover diary, written instructions on diary completion, and a pen. A trained research assistant will meet with the participant face to face or via telephone and explain how to use the diary. Instructions will include recommended frequency for writing (at least twice a week) and tips on how to express themselves. Potential topics will also be addressed, including what to write about in the beginning, during the ICU, and after ICU discharge. The hard copy of the diary will remain with the family member participant, and they will be asked to continue writing in the diary at least until patient discharge from the hospital. Research assistants will check in with participants via weekly telephone calls to provide prompts to remind them to use the diary and support, as needed, if the participant reports difficulty in writing diary entries. These calls will last approximately 1-5 minutes and will continue until patient discharge from the hospital.
  Other Names: Family-Authored ICU Diaries to Reduce Fear
  Arms: FAID Fear Intervention

SUMMARY:
The present study will:

Aim 1: Enroll 15 family members of CA patients to (a) pilot recruitment procedures, (b) estimate retention, and (c) assess acceptability of study procedures.

Family members will be randomized to either complete an ICU diary or to a control condition, and will complete surveys in the ICU, at patient discharge, and 30 days post-discharge.

Aim 2: Obtain an estimate of the association of intervention v. control with (i) family member fear (operationalized as cardiac anxiety about the patients' cardiac condition) at hospital discharge and (ii) family member PTSS 30 days post-discharge.

Exploratory Aims: Obtain an estimate of the association of intervention v. control with family member aversive cognitions towards exercise at hospital discharge.

DETAILED DESCRIPTION:
A cardiac arrest (CA) is a terrifying experience for patients, but maybe even more so for their loved ones. CA patients often have little to no memory of the CA and are often unconscious for substantial parts of their hospitalization, particularly their time in the intensive care unit (ICU) . In contrast, family members often witness all of these things, resulting in high levels of fear and psychological distress in family members. This phenomenon is so prevalent that it has been termed Post-Intensive Care Syndrome - Family (PICS - Family).

Critically, emotions are socially transmitted and memories are socially constructed. In this manner, family members can transmit their distress onto patients. Prior research has suggested that patients experiencing CA will develop memories of the CA event over time - potentially because they are trying to "fill in the gaps" in their memory. As such, family members may play a critical role in creating and cementing fear-based memories and distress in patients experiencing a CA. CA patients often report cardiac fear and preoccupation. This is not without consequence: fear-based distress, particularly early anxiety related to symptoms (e.g., rapid heartbeat) and markers for PTSS in other patient populations predicts reduced engagement in behavior necessary for secondary prevention (e.g., reduced physical activity) and increased morbidity and mortality. Distress in family members can also have an adverse impact on patients by undermining the capacity of family members to provide effective social support that can buffer patient distress.

A prior clinical trial found that family-authored diaries significantly reduced PTSS in family members (26.3% lower in intervention v. control conditions, 95% CI 4.8, 52.2) and trended towards a reduction in PTSS for patients (11.2% lower, 95% CI 15.7, 46.8). However, mechanisms of these effects were not examined, and no dyadic effects were tested. Furthermore, these previous diary studies have been conducted with the intention of sharing diaries with patients.

The present study will test the feasibility involving a similar Family-Authored ICU-diary intervention to reduce a proximal, dyadic mechanism: fear of CA in patients' family members. The target audience of the diary is thus family members, and patients will not see the diary unless the family member individually chooses to share it. The feasibility of targeting family member well-being alone is untested. The long-term goal is conducting a large scale randomized clinical trial (RCT) that tests whether a family-authored ICU diary can reduce fear of cardiac arrest in family members, and in turn, improve patients' mental wellbeing, health behaviors, and, ultimately, health outcomes.

ELIGIBILITY:
Inclusion Criteria

1. The family member of a patient who has experienced a cardiac arrest
2. Age 18 years and over
3. Able to speak, read, and write in English or Spanish
4. Participating in the CANOE study (AAAR8497) and indicated they were willing to hear about future research opportunities
5. Willing to write in a journal about their experiences

Exclusion Criteria

1. Unavailable for follow-up
2. Medical or psychiatric impairment that would prevent them from complying with the research protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Talea Cornelius, PhD, MSW, MS, Principal Investigator — Assistant Professor of Medicine
Locations (1):
- CUIMC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Explicit permission from participants to post de-identified data online was not obtained; rather, participants consented that, "Upon removal of identifiers from the dataset, data may be shared with other researchers." In accordance with recommendations for sharing raw clinical data for publication stating that it is ideal to obtain this consent, data are available only by request from the study PI.
  Hrynaszkiewicz I, Norton ML, Vickers AJ, Altman DG. Preparing raw clinical data for publication: guidance for journal editors, authors, and peer reviewers. Bmj. 2010;340.

REFERENCES:
- [Background] Davidson JE, Jones C, Bienvenu OJ. Family response to critical illness: postintensive care syndrome-family. Crit Care Med. 2012 Feb;40(2):618-24. doi: 10.1097/CCM.0b013e318236ebf9. PMID 22080636
- [Background] Gump BB, Kulik JA. Stress, affiliation, and emotional contagion. J Pers Soc Psychol. 1997 Feb;72(2):305-19. doi: 10.1037//0022-3514.72.2.305. PMID 9107002
- [Background] Rossignac-Milon M, Higgins ET. Epistemic companions: shared reality development in close relationships. Curr Opin Psychol. 2018 Oct;23:66-71. doi: 10.1016/j.copsyc.2018.01.001. Epub 2018 Jan 11. PMID 29360060
- [Background] French CC. Dying to know the truth: visions of a dying brain, or false memories? Lancet. 2001 Dec 15;358(9298):2010-1. doi: 10.1016/S0140-6736(01)07133-1. No abstract available. PMID 11755600
- [Background] Rosman L, Whited A, Lampert R, Mosesso VN, Lawless C, Sears SF. Cardiac anxiety after sudden cardiac arrest: Severity, predictors and clinical implications. Int J Cardiol. 2015 Feb 15;181:73-6. doi: 10.1016/j.ijcard.2014.11.115. Epub 2014 Nov 18. PMID 25482282
- [Background] Edmondson D, Richardson S, Falzon L, Davidson KW, Mills MA, Neria Y. Posttraumatic stress disorder prevalence and risk of recurrence in acute coronary syndrome patients: a meta-analytic review. PLoS One. 2012;7(6):e38915. doi: 10.1371/journal.pone.0038915. Epub 2012 Jun 20. PMID 22745687
- [Background] Monane R, Sanchez GJ, Kronish IM, Edmondson D, Diaz KM. Post-traumatic stress disorder symptoms and aversive cognitions regarding physical activity in patients evaluated for acute coronary syndrome. Eur J Prev Cardiol. 2018 Mar;25(4):402-403. doi: 10.1177/2047487317746255. Epub 2017 Dec 4. No abstract available. PMID 29198138
- [Background] Rafaeli E, Gleason ME. Skilled support within intimate relationships. Journal of Family Theory & Review. 2009;1(1):20-37.
- [Background] Nielsen AH, Angel S, Egerod I, Hansen TB. The effect of diaries written by relatives for intensive care patients on posttraumatic stress (DRIP study): protocol for a randomized controlled trial and mixed methods study. BMC Nurs. 2018 Aug 16;17:37. doi: 10.1186/s12912-018-0306-y. eCollection 2018. PMID 30127664
- [Background] Nielsen AH, Angel S, Egerod I, Lund TH, Renberg M, Hansen TB. The effect of family-authored diaries on posttraumatic stress disorder in intensive care unit patients and their relatives: A randomised controlled trial (DRIP-study). Aust Crit Care. 2020 Mar;33(2):123-129. doi: 10.1016/j.aucc.2019.01.004. Epub 2019 Feb 20. PMID 30795978

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant enrolled on November 29, 2021, and the last enrolled on September 30, 2022. Follow-up sessions occurred between January 21, 2022-November 30, 2022.
Pre-assignment Details: The baseline/pre-intervention session was conducted in person or over the telephone. During the baseline/pre-intervention session, participants (1) provided verbal consent, (2) were randomized, and (3) completed baseline assessments.
Period: Overall Study
Arm/Group | FAID Fear Intervention | Control Condition - Usual Care
Started | 11 | 5
Completed | 10 | 4
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: One participant in the FAID Fear Intervention withdrew immediately after randomization, prior to completing baseline demographic assessments.
Groups:
- Total: Total of all reporting groups
Arm/Group | FAID Fear Intervention | Control Condition - Usual Care | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.50 (13.32) | 49.20 (15.04) | 50.73 (13.41)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Woman | 9 | 3 | 12
  Gender: Man | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 8 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 15
Language [Count of Participants; unit: Participants]
  English | 8 | 4 | 12
  Spanish | 2 | 1 | 3
Health Insurance [Count of Participants; unit: Participants]
  Yes | 8 | 5 | 13
  No | 2 | 0 | 2
Education [Count of Participants; unit: Participants]
  No Formal Education | 0 | 0 | 0
  Less than High School | 0 | 0 | 0
  Some High School | 0 | 0 | 0
  High School/GED | 2 | 2 | 4
  Trade/Vocational School | 0 | 0 | 0
  Some College | 2 | 1 | 3
  Associate's Degree | 1 | 0 | 1
  College Degree | 3 | 1 | 4
  Graduate/ Professional Degree | 2 | 1 | 3
Income [Count of Participants; unit: Participants] — Population: This question was added partway through the study.
  Participants
    number analyzed (Participants) | 6 | 3 | 9
    $0 | 0 | 0 | 0
    $1 - $9,999 | 0 | 0 | 0
    $10,000 - $24,999 | 2 | 0 | 2
    $25,000 - $49,999 | 2 | 1 | 3
    $50,000 - $74,999 | 0 | 0 | 0
    $75,000 - $99,999 | 0 | 0 | 0
    $100,000 - $149,999 | 1 | 0 | 1
    $150,000 or more | 1 | 0 | 1
    Decline to Respond | 0 | 2 | 2
Relationship to Patient [Count of Participants; unit: Participants]
  Partner | 7 | 3 | 10
  Child | 2 | 1 | 3
  Parent | 1 | 0 | 1
  Sibling | 0 | 1 | 1
Live with Patient [Count of Participants; unit: Participants]
  Yes | 9 | 4 | 13
  No | 1 | 1 | 2
Relationship Length (Partners of Patients Only) [Mean (Standard Deviation); unit: years] — Population: This was reported by partner of patients only.
  years
    number analyzed (Participants) | 7 | 3 | 10
    (all) | 19.86 (11.77) | 22.67 (19.14) | 20.70 (13.25)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eligible Family Members of Cardiac Arrest (CA) Patients Who Agree/Consent to Participate in the Pilot Study
Description: This is to assess feasibility of recruitment. Potential family member participants whom the study team approaches and agree/consent to take part in the study will be tallied.
  Specifically, we divided the number of family member participants who enrolled in the study by the number of potential participants referred to the study (enrolled/referred).
Time Frame: Baseline (ICU admittance)
Measure: Count of Participants; unit: Participants
Groups:
- All Referrals to FAID Fear: 25 potential participants met preliminary eligibility and were referred to study staff for recruitment.
  Participants were recruited from among those who were enrolled in the Cardiac Neuropsychosocial Outcomes Evaluation - Family (CANOE-F; R01 HL153311; PI Agarwal) substudy, an observational cohort study of family members of CA patients within CUIMC/NewYork-Presbyterian Hospital (NYPH). Only CANOE-F participants who enrolled while the patient was still in the ICU and who agreed to be contacted about future research opportunities were approached for participation in this study.
  Participant eligibility criteria additionally included (1) primary partner or family member of a patient who was hospitalized at CUIMC for a CA, (2) age 18 years or over, (3) able to speak, read, and write in English or Spanish, (4) willing to write in a journal about their experiences, and (5) available for follow-up. Participants were excluded if they presented any medical or psychiatric impairment that would have prevented them from complying with the research protocol.
Arm/Group | All Referrals to FAID Fear
Number analyzed (Participants) | 25
Participants
  Agreed to Participate | 16
  Declined to Participate | 4
  Unable to Reach | 5
Statistical Analysis 1: Comparison: All Referrals to FAID Fear; Test type: Other — Proportion of referrals who provided consent and enrolled into the study was calculated; Proportion = 0.640, 95% CI 2-sided [0.425 to 0.820]

2. Primary Outcome: Proportion of Enrolled Family Members Who Complete the Pilot Study
Description: This is to estimate/assess retention. Family members who remain in the study at the final assessment will be tallied.
  Specifically, we divided the number of family member participants who completed the study by the number of potential participants who did not complete the study (completed/did not complete).
Time Frame: 30 days post-discharge
Population: Proportion of enrolled participants who remained in the study 30 days after the end of hospital care was calculated.
Measure: Count of Participants; unit: Participants
Groups:
- All FAID Fear Enrollments: All participants enrolled in FAID Fear (intervention and control)
Arm/Group | All FAID Fear Enrollments
Number analyzed (Participants) | 16
Participants
  Remained in FAID Fear | 14
  Withdrew from FAID Fear | 2
Statistical Analysis 1: Comparison: All FAID Fear Enrollments; Test type: Other — Proportion of enrolled participants who remained in the study at 30 days after the end of hospital care was calculated; Proportion = 0.875, 95% CI 2-sided [0.617 to 0.985]

3. Secondary Outcome: Proportion of Family Members That Adhere to the Diary Intervention
Description: This is to assess acceptability of study procedures. Family members who report completing at least 2 diary entries/week will be tallied.
  Specifically, we divided the number of family member participants in the diary intervention who adhered to the intervention by the number of participants who did not adhere to the intervention (adhered/did not adhere).
Time Frame: Up to hospital discharge (approximately 21 days)
Measure: Count of Participants; unit: Participants
Arm/Group | FAID Fear Intervention
Number analyzed (Participants) | 11
Participants
  Adherent to Diary Intervention | 7
  Not Adherent to Diary Intervention | 4
Statistical Analysis 1: Comparison: FAID Fear Intervention; Test type: Other — Proportion of participants randomized to the FAID Fear Diary Intervention who wrote in the diary at least twice per week up until the end of hospital care was calculated; Proportion = 0.636, 95% CI 2-sided [0.308 to 0.891]

4. Secondary Outcome: Proportion of Family Members That Complete the Majority of Survey Assessments
Description: This is to assess acceptability of study procedures. Family members who complete at least 90% of survey assessments will be tallied.
  Specifically, we divided the number of family member participants who completed at least 90% of survey assessments by the number of family member participants who completed less than 90% of survey assessments (completed/did not complete).
Time Frame: Up to 30 days post-discharge
Measure: Count of Participants; unit: Participants
Arm/Group | All FAID Fear Enrollments
Number analyzed (Participants) | 16
Participants
  Provided Data for >= 90% of Assessments | 14
  Provided Data for < 90% of Assessments | 2
Statistical Analysis 1: Comparison: All FAID Fear Enrollments; Test type: Other — Proportion of enrolled participants who provided complete data for at least 90% of all study assessments was calculated; Proportion = 0.875, 95% CI 2-sided [0.617 to 0.985]

5. Secondary Outcome: Proportion of Family Members That Agree That the Intervention Was Acceptable
Description: As a measure of intervention acceptability, study will assess the proportion of participants who agree that the intervention was acceptable for reducing cardiac anxiety about the patient's heart using mean of the 4-item Acceptability of Intervention Measure (score >= 4; 1 = completely disagree, 5 = completely agree). Possible mean scores range from 1 to 5.
  Specifically, we divided the number of family member participants in the diary intervention who agreed the intervention was acceptable by the number of family member participants in the diary intervention who did not agree that the intervention was acceptable (acceptable/not acceptable).
Time Frame: 30 days post-discharge
Population: Excludes participant who withdrew immediately following randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | FAID Fear Intervention
Number analyzed (Participants) | 10
Participants
  Acceptable | 8
  Not Acceptable | 2
Statistical Analysis 1: Comparison: FAID Fear Intervention; Test type: Other — Proportion of intervention participants who agreed that the ICU diary was acceptable for reducing fear about their loved one's heart was calculated; Proportion = 0.800, 95% CI 2-sided [0.444 to 0.975]

6. Secondary Outcome: Proportion of Family Members That Agree That the Intervention Was Feasible
Description: As a measure of intervention acceptability, study will assess the proportion of participants who agree that the study was feasible using the mean of the 4-item Feasibility of Intervention Measure (score >= 4; 1 = completely disagree, 5 = completely agree). Possible mean scores range from 1 to 5.
  Specifically, we divided the number of family member participants in the diary intervention who agreed the intervention was feasible by the number of family member participants in the diary intervention who did not agree that the intervention was feasible (feasible/not feasible).
Time Frame: 30 days post-discharge
Population: Excludes one participant who withdrew immediately after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | FAID Fear Intervention
Number analyzed (Participants) | 10
Participants
  Feasible | 9
  Not Feasible | 1
Statistical Analysis 1: Comparison: FAID Fear Intervention; Test type: Other — Proportion of intervention participants who agreed that the ICU diary was feasible for reducing fear about their loved one's heart was calculated; Proportion = 0.900, 95% CI 2-sided [0.555 to 0.998]

7. Secondary Outcome: Proportion of Family Members That Agree That the Intervention Was Appropriate
Description: As a measure of intervention acceptability, study will assess the proportion of participants who agree that the study was appropriate for reducing cardiac anxiety about the patient's heart using the 4-item Intervention Appropriateness Measure (score >= 4; 1 = completely disagree, 5 = completely agree). Possible mean scores range from 1 to 5.
  Specifically, we divided the number of family member participants in the diary intervention who agreed the intervention was appropriate by the number of family member participants in the diary intervention who did not agree that the intervention was appropriate (appropriate/not appropriate).
Time Frame: 30 days post-discharge
Population: Excludes one participant who withdrew immediately following randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | FAID Fear Intervention
Number analyzed (Participants) | 10
Participants
  Appropriate | 7
  Not Appropriate | 3
Statistical Analysis 1: Comparison: FAID Fear Intervention; Test type: Other — Proportion of intervention participants who agreed that the ICU diary was appropriate for reducing fear about their loved one's heart was calculated; Proportion = 0.700, 95% CI 2-sided [0.348 to 0.933]

8. Other Pre Specified Outcome: Cardiac Anxiety Questionnaire Fear Subscale Score
Description: This is to measure family members' cardiac anxiety about the patients' heart. Cardiac anxiety will be measured using the 8-item fear subscale of the Cardiac Anxiety Questionnaire and compared between intervention and control participants (higher scores indicate greater fear; 1 = never, 5 = always). Possible mean scores range from 1 to 5.
Time Frame: Hospital discharge (approximately 21 days), 30 days post-discharge
Population: Excludes two participants who withdrew before completing assessments at the end of hospital care.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAID Fear Intervention | Control Condition - Usual Care
Number analyzed (Participants) | 10 | 4
score on a scale
  End of Hospital Care | 3.35 (0.90) | 3.59 (0.61)
  30 Days After End of Hospital Care | 3.33 (0.88) | 3.41 (0.33)
Statistical Analysis 1: Comparison: FAID Fear Intervention vs Control Condition - Usual Care; Outcome analysis at the end of hospital care; Test type: Superiority; p = .63, t-test, 2 sided; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.83 to 1.32]
Statistical Analysis 2: Comparison: FAID Fear Intervention vs Control Condition - Usual Care; Outcome analysis for 30 days after the end of hospital care; Test type: Superiority; p = .86, t-test, 2 sided; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.92 to 1.08]

9. Other Pre Specified Outcome: Cardiac Anxiety Questionnaire Avoidance Subscale Score
Description: This is to measure family members' aversive cognitions towards patients' exercise. Aversive cognitions towards exercise will be measured using the 5-item avoidance subscale of the Cardiac Anxiety Questionnaire and compared between intervention and control participants (higher scores indicate greater aversive cognitions; 1 = never, 5 = always). Possible mean scores range from 1 to 5.
Time Frame: Hospital discharge (approximately 21 days), 30 days post-discharge
Population: Excludes two participants who did not provide data for these assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAID Fear Intervention | Control Condition - Usual Care
Number analyzed (Participants) | 10 | 4
score on a scale
  End of Hospital Care | 3.56 (1.14) | 3.45 (0.53)
  30 Days After End of Hospital Care | 3.16 (1.07) | 3.35 (0.72)
Statistical Analysis 1: Comparison: FAID Fear Intervention vs Control Condition - Usual Care; Outcome analysis for the end of hospital care; Test type: Superiority; p = .86, t-test, 2 sided; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-1.43 to 1.21]
Statistical Analysis 2: Comparison: FAID Fear Intervention vs Control Condition - Usual Care; Outcome analysis for 30 days after the end of hospital care; Test type: Superiority; p = .75, t-test, 2 sided; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-1.10 to 1.58]

10. Other Pre Specified Outcome: Posttraumatic Stress Disorder Checklist Score
Description: This is to measure family members' posttraumatic stress symptoms in relation to the patients' cardiac arrest at discharge. Posttraumatic stress symptoms will be measured using the sum of the 20-item Posttraumatic Stress Disorder Checklist cued to the CA-event and related hospitalization and compared between intervention and control participants. A score >=33 is considered a positive screen for PTSD (higher scores indicate greater PTSD symptoms; 0 = not at all, 4 = extremely). Possible total scores range from 0 to 80.
Time Frame: 30 days post-discharge
Population: Excludes two participants who did not provide data for this assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAID Fear Intervention | Control Condition - Usual Care
Number analyzed (Participants) | 10 | 4
score on a scale | 19.70 (12.83) | 11.00 (4.08)
Statistical Analysis 1: Comparison: FAID Fear Intervention vs Control Condition - Usual Care; Test type: Superiority; p = .22, t-test, 2 sided; Mean Difference (Final Values) = -8.70, 95% CI 2-sided [-23.26 to 5.86]
Statistical Analysis 2: Comparison: FAID Fear Intervention vs Control Condition - Usual Care; Test type: Superiority; p = .26, Wilcoxon (Mann-Whitney); χ2(1) = 1.29
Statistical Analysis 3: Comparison: FAID Fear Intervention vs Control Condition - Usual Care; A Fisher's Exact Test was conducted to compare the number of participants with a positive screen for PTSD symptoms (score >=33) to those who did not have a positive screen for PTSD symptoms (score < 33); Test type: Superiority; p = 1.00, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from baseline enrollment through the final assessment. For participants who completed the study this monitoring period ranged from 34 days to 151 days (Median = 46 days). For the two participants who completed the study, monitoring lasted for 0 days (one individual dropped out immediately after random assignment, the other dropped out when contacted at the end of hospital care and did not report any data/complete any assessments at this time).
Arm/Group | FAID Fear Intervention | Control Condition - Usual Care
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT05144477/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT05144477/SAP_001.pdf